CLINICAL TRIAL: NCT05592665
Title: PRO-VISION: Patient Reported Outcomes-Based Monitoring of VEGF-Inhibitor Side Effects in ONcology
Acronym: PRO-VISION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2126
Record Dates: First submitted 2022-09-20; First posted 2022-10-25 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Renal Cell Carcinoma
Keywords: patient reported outcomes; vascular endothelial growth factor; quality of life; adverse effects
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Perspective (Other): Study participants will complete several questionnaires/assessments related to adverse events and quality of life.
  Interventions: Other: Survey Questionnaire

INTERVENTIONS:
Other: Survey Questionnaire — Study participants will complete several questionnaires/assessments via PRO-Core standardized email communication or via telephone with a study team member.

SUMMARY:
The purpose of this study is to investigate how collecting information about treatment-related side effects directly from patients can help manage the side effects associated with certain oral chemotherapies. This study is specifically investigating this approach in patients taking oral vascular endothelial growth factor receptor (VEGFR) tyrosine kinase inhibitors (TKIs) for metastatic renal cell carcinoma (mRCC).

Participants in this study will receive a survey via email or telephone once a week while receiving treatment with a VEGFR TKI. The survey will ask about symptoms such as nausea or fatigue and overall quality of life. This survey should take no more than 15 minutes to complete.

The survey will be sent directly to the oncology care team. Participants will receive a follow-up phone call or message from the team when participants have new or worsening symptoms. The participants will continue to receive surveys for as long as they are receiving a VEGF TKI treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older
* Histologically confirmed renal cell carcinoma requiring treatment with VEGF TKI.
* Patients may be receiving other concurrent cancer-directed therapy such as immune checkpoint inhibitors.
* English or Spanish speaking
* Ability to complete PRO surveys (i.e. ability to read/write or access to telephone or internet)
* Willing and able to meet all study requirements

Exclusion Criteria:

All subjects meeting any of the exclusion criteria at baseline will be excluded from study participation.

• Inability for any reason to complete PRO surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2027-01-16 (Estimated); Study Completion 2031-01-16 (Estimated)

PRIMARY OUTCOMES:
Relative dose intensity | Up to 3 years
  Relative dose intensity is defined as the actual treatment dose taken per unit of time divided by the standard or initially prescribed dose per unit during the duration of treatment with VEGF TKI.

SECONDARY OUTCOMES:
Dose modifications | Up to 3 years
  The proportion of patients who change the dose of VEGF TKI study treatment during the duration of treatment with VEGF TKI therapy.
Dose interruption | Up to 3 years
  The proportion of patients who change the dose of VEGF TKI study treatment during the duration of treatment with VEGF TKI therapy.
Hospital admissions | Up to 3 years
  The proportion of patients requiring hospitalization for a treatment-related side effect.
Emergency department visits | Up to 3 years
  The proportion of patients requiring an emergency department visit for treatment-related adverse events.
Duration of treatment on initial VEGF TKI dose | Up to 3 years
  Duration of treatment on initial VEGF TKI dose is defined from day 1 of treatment until the first dose reduction or dose interruption.
Duration of treatment on VEGF TKI regimen | Up to 3 years
  Duration of treatment on VEGF TKI regimen is defined from day 1 of treatment until the last dose of VEGF TKI treatment at any dose.
Progression-free survival | Up to 3 years
  Progression-free survival is defined as day 1 of treatment until progression of disease or death from any cause; patients will be censored at the time of new treatment initiation if progression has not occurred.
Health-related quality of life and symptom burden -Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events | Up to 3 years
  Health-related quality of life (HRQoL) and symptom burden will be assessed using the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) questionnaire.
  The PRO-CTCAE Measurement System characterizes the frequency, severity, interference, and presence/absence of symptomatic toxicities that include pain, fatigue, nausea, and cutaneous side effects such as rash and hand-foot syndrome, all toxicities that can be meaningfully reported from the patient perspective.
Health-related quality of life and symptom burden - EuroQol-5 Dimension (EQ-5D-5L) questionnaire. | Up to 3 years
  Health-related quality of life (HRQoL) and symptom burden will be assessed using the EuroQol-5 Dimension (EQ-5D-5L) questionnaire.
  The EQ-5D-5L is a QoL assessment that comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels ranging from no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5) to extreme problems.
Health-related quality of life and symptom burden- Functional Assessment of Cancer Therapy Kidney System Index | Up to 3 years
  Health-related quality of life (HRQoL) and symptom burden will be assessed using the Functional Assessment of Cancer Therapy Kidney System Index (FKSI-19) scores.
  The FKSI-19 is a 19-item questionnaire specific to kidney cancer. The items include disease-related symptoms(both physical and emotional), as well as treatment side-effects, and function/well-being. The questions are reported on a Likert scale as not at all, a little bit, somewhat, quite a bit, or very much. The questions address lack of energy, pain, weight loss, fatigue, shortness of breath, fevers, bone pain, cough, weakness, blood in urine, appetite, sleep, worry about the condition, nausea, diarrhea, bothered by side effects, ability to work, ability to enjoy life and level of content with the quality of life.
Treatment satisfaction | Up to 3 years
  The proportion of subjects satisfied or very satisfied with the weekly surveys to help manage side effects.
VEGF TKI treatment adherence | Up to 3 years
  The median number of doses missed in a 4-week treatment period.
Adherence to Patient Reported Outcome -based symptom | Up to 3 years
  Adherence to Patient Reported Outcome (PRO)-based symptom monitoring will be defined as the proportion of surveys completed per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Rose, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.

REFERENCES:
- See also: Related Info — http://unclineberger.org/patientcare/clinical-trials/clinical-trials